CLINICAL TRIAL: NCT07082374
Title: Dual Subsartorial Block Versus Adductor Canal Block Versus Femoral Nerve Block for Postoperative Analgesia in Patients Undergoing Total Knee Arthroplasty: A Randomized Clinical Trial
Brief Title: Dual Subsartorial Versus Adductor Canal Block Versus Femoral Nerve Block for Postoperative Analgesia in Patients Undergoing Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1260/6/25
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Dual Subsartorial Block; Adductor Canal Block; Femoral Nerve Block; Postoperative Analgesia; Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DSB group (Experimental): Patients will receive dual subsartorial block (DSB).
  Interventions: Other: Dual subsartorial block
- ACB group (Experimental): Patients will receive an adductor canal block (ACB).
  Interventions: Other: Adductor canal block
- FNB group (Experimental): Patients will receive a femoral nerve block (FNB).
  Interventions: Other: Femoral nerve block

INTERVENTIONS:
Other: Dual subsartorial block — Patients will receive dual subsartorial block (DSB).
  Arms: DSB group
Other: Adductor canal block — Patients will receive an adductor canal block (ACB).
  Arms: ACB group
Other: Femoral nerve block — Patients will receive a femoral nerve block (FNB).
  Arms: FNB group

SUMMARY:
This study aims to compare the effect of dual subsartorial block (DSB), adductor canal block (ACB), and femoral nerve block (FNB) for postoperative analgesia in patients undergoing total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) offers increased joint mobility and painless ambulation to patients. Femoral nerve block (FNB) is commonly used to relieve postoperative pain and opioid consumption.

Adductor canal block (ACB) is a common analgesic intervention for postoperative pain control following TKA. The dual subsartorial block (DSB) is a novel procedure-specific and motor-sparing regional analgesia (RA) technique that may reduce overall postoperative opioid consumption when used in conjunction with multimodal analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Undergoing total knee arthroplasty (TKA) under general anesthesia.

Exclusion Criteria:

* Severe valgus deformity.
* Acute/chronic kidney disease.
* Neurological deficit.
* Cognitive dysfunction.
* Local infection at the site of injection.
* Coagulopathy.
* Hypersensitivity and/or allergies to local anesthetic (LA) or any of the study medications.
* Chronic opioid consumption (daily or almost daily use of opioids for > three months).
* Operative limb neuropathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery to first dose of morphine administrated).

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the visual analog scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at PACU, 2, 4, 6, 8, 12, 18 and 24 h postoperatively.
Degree of patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, pruritus, or any other complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.